CLINICAL TRIAL: NCT01204983
Title: Quality Improvement Project - Evaluation of Current Standard of Care for Feeding Practices With Donor Human Milk Products in the NICU
Brief Title: Quality Improvement Project - Evaluation of Current Standard of Care for Feeding Practices in the NICU
Acronym: NICU
Status: Completed | Type: Observational
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Amy Hair, Assistant Professor, Baylor College of Medicine
Other Study IDs: H-26923
Record Dates: First submitted 2010-09-16; First posted 2010-09-20 (Estimated); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Infant, Very Low Birth Weight
Keywords: very low birth weight infant; donor human milk

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observational: This is a quality improvement project to evaluate the current standard of care of nutritional management for very low birth weight infants receiving donor human milk products in the NICU at Texas Children's Hospital.
  There is no randomization, there are no control subjects, and therefore there is no probability of group assignment.

SUMMARY:
Human milk is associated with substantial benefits to infants' health and development, especially in premature infants. Some mothers are unable or unwilling to provide breast milk to their infant. The use of donor human milk as an alternative to cow milk in these infants has risen dramatically in the past year. However, there have been recent reports of hyperphosphatemia and hyponatremia associated with the consumption of donor human milk products. These electrolyte imbalances can lead to concerning symptoms, including headache, nausea, vomiting, altered mental status, coma, seizures, or heart failure. It is important to recognize and appropriately treat these electrolyte disturbances associated with donor human milk to avoid potential nutritional problems.

DETAILED DESCRIPTION:
This is a quality improvement project to evaluate the current standard of care of nutritional management for very low birth weight infants receiving donor human milk products in the NICU at Texas Children's Hospital.

There is no randomization, there are no control subjects, and therefore there is no probability of group assignment.

Infants will be identified by the dietitian staff at TCH upon admission to the NICU (Levels 2 and 3) and communicated to the PI and PI's staff.

For each subject, data collection will begin at the point that the infant first receives any enteral feeding (including trophic feeds). All infants less than or equal to 1250 g birth weight will be followed initially. If the parent declines to allow donor human milk products for the infant, this will be noted in the data collection and no additional data will be collected for this infant. If at a later time, the parent decides to allow donor human milk products, we will begin data collection again. Our current experience is that >95% of mothers agree to donor human milk products.

Data collection will continue throughout the hospitalization until one week after all donor human milk products have been discontinued or discharge.

From the medical chart, we will record the following data on a weekly basis: weight, length, head circumference, labs (Chem 10 panel - BUN, creatinine, sodium, potassium, bicarbonate, chloride, calcium, phosphorus, magnesium, and glucose), medications, and the nutrition order (parenteral and enteral nutrition feeding orders including volume, concentration, and additives). If an abnormal nutrition-related lab is noted, changes in the nutrition order will be recorded more frequently than on a weekly basis. A copy of the data collection template is attached in Section S.

No labs will be requested for research purposes. No interventions are part of this protocol. This protocol involves only minimal risk to individuals. A waiver of consent would not in any way adversely affect the privacy rights and the welfare of the individuals.

ELIGIBILITY:
Inclusion Criteria:

* Premature infants (<37 weeks gestation) with a birth weight less than or equal to 1250 grams.

Exclusion Criteria:

* Infants with a birth weight greater than 1250 grams
* Infants transferred from an outside hospital to TCH at greater than 21 days of age
* Infants who do not achieve any enteral feeds by 4 weeks of age
* Infants with major congenital anomalies

Min Age: 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Premature, very low birth weight infants only
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2010-07-01 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
To evaluate the current standard of care of nutritional management | August 2010 - December 2011
  To evaluate the current standard of care of nutritional management for very low birth weight infants receiving donor human milk products in the NICU at Texas Children's Hospital.

SECONDARY OUTCOMES:
To ensure that guidelines for VLBW infants are followed | August 2010 - December 2011
  To ensure that guidelines to monitor electrolytes in infants < 1250 g receiving donor human milk products are being followed and that appropriate interventions are being given if abnormalities are determined.

CONTACTS AND LOCATIONS:
Overall Officials: Amy Hair, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine / Texas Children's Hospital, Houston, Texas, United States